CLINICAL TRIAL: NCT00075283
Title: Gait Restoration In Hemiparetic Stroke Patients Using Goal-Directed, Robotic-Assisted, Treadmill Training
Brief Title: Walking Therapy In Hemiparetic Stroke Patients Using Robotic-Assisted Treadmill Training
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: U.S. Department of Education (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H133E020724; IRB 2002-427
Record Dates: First submitted 2004-01-08; First posted 2004-01-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Hemiparesis; Stroke
Keywords: Physical Therapy; Locomotion therapy; Gait training; Stroke; Robotics; Rehabilitation; Treadmill; Hemiparetic stroke; Unilateral brain lesion
MeSH Terms: conditions — Paresis; Stroke

INTERVENTIONS:
Device: Lokomat (Robotic Orthosis) combined with slat belt treadmill

SUMMARY:
The overall goal of this study is to determine whether robotic-assisted gait training is better than standard physical therapy treatments for improving walking ability in hemiparetic stroke patients.

DETAILED DESCRIPTION:
Subjects enrolled into the study will be randomly assigned to one of 2 groups. The first group will receive one hour of conventional gait training, consisting of lower extremity strengthening exercises, stretching, and full weight bearing walking as tolerated, with appropriate physical assistance from a therapist. The second group will receive walking therapy using a Lokomat, which is a special treadmill that works in conjunction with 2 light-weight robotic arms that assists the subject to move their legs while they try to walk on the treadmill. Some of the subject's body-weight will be supported using a harness. During Lokomat training sessions, subjects will receive feedback of their walking performance on a computer monitor to help them walk. Both groups will be trained for 8-10 weeks, 3 times per week, for 1 hour training sessions (24 total sessions). Resources for transportation to the National Rehabilitation Hospital will be provided to all study participants.

ELIGIBILITY:
Inclusion:

* Unilateral brain lesion.
* Within 6 months post-stroke.
* Receiving no other therapy targeting function of lower limb.
* Demonstration of hemiparesis (motor dysfunction in lower limb).
* Able to walk 5 meters without therapist assistance (walking device only).
* Able to follow commands and protocol.

Exclusion:

* Significant cognitive or communication impairments.
* Uncontrolled hypertension.
* Uncontrolled diabetes.
* Clinical depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-11

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joseph M Hidler, Ph.D., Principal Investigator — The Catholic University of America
Locations (1):
- National Rehabilitation Hospital, Washington D.C., District of Columbia, United States